CLINICAL TRIAL: NCT00005388
Title: Visceral Fat, Metabolic Rate, and CHD Risk in Young Adults
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4294; R01HL053359 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2004-04

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Disease; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Coronary Disease; Obesity

SUMMARY:
To measure visceral (intraabdominal) fat by computerized tomography (CT) scan and to measure resting metabolic rate by indirect calorimetry in 400 CARDIA subjects, ages 28-40 years (100 of each race/gender group) from the Oakland, California and Birmingham, Alabama centers.

DETAILED DESCRIPTION:
BACKGROUND:

The prevalence of obesity increased markedly in the United States from the 1960's to the 1980's, and varied by race and gender with particularly high rates of obesity among Black women. Reasons for the ethnic differences in the prevalence of obesity were not understood. This cross-sectional study was performed in conjunction with the 10-year follow-up examination for the Coronary Artery Risk Development in Young Adults (CARDIA) study, an NHLBI-funded longitudinal study of development of risk factors for coronary heart disease (CHD) in young black and white adults.

This study represented a unique opportunity to investigate factors that may influence the development of obesity, to better understand the relationship between obesity and cardiovascular risk factors, and to increase understanding of racial differences in adiposity.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

DESIGN NARRATIVE:

The cross-sectional study tested the hypothesis that visceral adipose tissue, the component of fat considered to be most strongly related to coronary heart disease (CHD) risk factors, differed in Black and white subjects. Specifically, the investigators proposed that Black subjects had less visceral adipose tissue for a given level of total body fat than white subjects. Further, the relationship between visceral adipose tissue and risk factors for CHD was similar in all subjects. This would explain the different relationship between obesity and CHD risk factors seen in Black vs white subjects. A second specific aim was to determine whether Black women had a lower resting energy expenditure than Black men or whites. This could explain the higher prevalence of obesity in Black women than in Black men or whites of either gender. CT scans were recorded on tape and shipped to the University of Colorado Health Sciences Center where visceral adipose tissue was quantified. Dietary intake and physical activity were measured as important covariates in the relationship between metabolic rate and adiposity, and thyroid function was measured as a determinant of resting energy expenditure. The CARDIA study provided funding for cardiovascular risk factor measurements, including blood pressure, lipids, insulin, glucose, smoking, and anthropometric measurements including dual energy absorptiometry (DEXA) measurements of total and regional body fat.

The study was renewed in 1999 through March 2004 to perform a five-year follow-up of the cohort.

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1995-09; Study Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Sidney — Kaiser Foundation

REFERENCES:
- [Background] Sidney S, Lewis CE, Hill JO, Quesenberry CP Jr, Stamm ER, Scherzinger A, Tolan K, Ettinger B. Association of total and central adiposity measures with fasting insulin in a biracial population of young adults with normal glucose tolerance: the CARDIA study. Obes Res. 1999 May;7(3):265-72. doi: 10.1002/j.1550-8528.1999.tb00405.x. PMID 10348497
- [Background] Hill JO, Sidney S, Lewis CE, Tolan K, Scherzinger AL, Stamm ER. Racial differences in amounts of visceral adipose tissue in young adults: the CARDIA (Coronary Artery Risk Development in Young Adults) study. Am J Clin Nutr. 1999 Mar;69(3):381-7. doi: 10.1093/ajcn/69.3.381. PMID 10075320
- [Background] Sharp TA, Bell ML, Grunwald GK, Schmitz KH, Sidney S, Lewis CE, Tolan K, Hill JO. Differences in resting metabolic rate between white and African-American young adults. Obes Res. 2002 Aug;10(8):726-32. doi: 10.1038/oby.2002.99. PMID 12181380
- [Background] Simon JA, Murtaugh MA, Gross MD, Loria CM, Hulley SB, Jacobs DR Jr. Relation of ascorbic acid to coronary artery calcium: the Coronary Artery Risk Development in Young Adults Study. Am J Epidemiol. 2004 Mar 15;159(6):581-8. doi: 10.1093/aje/kwh079. PMID 15003962